CLINICAL TRIAL: NCT04526756
Title: Mechanical Thrombectomy for Acute Large Vessel Occlusion Stroke With Mild Symptoms After Imaging Selection
Brief Title: Mechanical Thrombectomy for Acute Large Vessel Occlusion Stroke With Mild Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-DFNE-002
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Ischemic Stroke; Acute Stroke
Keywords: acute ischemic stroke; acute large vessel occlusion; thrombectomy; mild stroke;; prognosis
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, controlled, outcome-blinded study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): patients in this group will receive mechanical thrombectomy and standardized drug treatment of acute ischemic stroke
  Interventions: Procedure: Mechanical Thrombectomy
- control group (No Intervention): patients in this group will receive standardized drug treatment of acute ischemic stroke

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — Solitaire stent and manual aspiration thrombectomy were performed as the first-line endovascular treatment
  Arms: Intervention group

SUMMARY:
Mechanical thrombectomy(MT) has been recommended in patients with acute large vessel occlusion stroke(LVO) , especially for those with National Institutes of Health Stroke Scale (NIHSS) score ≥6. However, it is still unclear if patients with minor strokes and LVO also benefit from MT.The aim of this study was to evaluate the safety and efficacy of MT for acute LVO and mild symptoms.

DETAILED DESCRIPTION:
This is a prospective cohort study of patients with with mild ischemic stroke (NIHSS Score <6) and LVO. Patients were divided into 2 groups: MT or medical management.Baseline data and clinical outcomes were compared. A independent clinical outcome was defined as a modified Rankin Scale score of 0 to 2 at 90 days. A excellent clinical outcome was defined as a modified Rankin Scale score of 0 to 1 at 90 days. Symptomatic intracranial hemorrhage(sICH) was the safety outcome.

ELIGIBILITY:
Inclusion Criteria:

1. acute ischemic stroke within 24 hours of symptom onset presenting cortical symptoms (such as aphasia, somnolence,slow-minded,etc.) or vertigo with bilateral pathological signs;
2. age≥18 years old;
3. the NIHSS score before evaluation of thrombectomy<6;
4. large artery occlusion including Middle cerebral artery M1, proximal M2 segment, intracranial internal carotid artery and infarct core volume≤50ml and mismatch ratio>1.8 or basilar artery and posterior cerebral artery P1 occlusion

Exclusion Criteria:

1. Patients without prior functional independence (mRS score of >2)
2. Patients in intervention group with occlusive artery spontaneous recanalization in digital subtraction angiography
3. patients in control group with neurological worsening and received rescue thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale(mRS) score of 0 to 2 | 90 days
  independent outcome at 90 days

SECONDARY OUTCOMES:
modified Rankin Scale(mRS) score of 0 to 1 | 90 days
  excellent outcome at 90 days

OTHER OUTCOMES:
Symptomatic intracranial haemorrhage transformation | 36 hours
  Symptomatic intracranial haemorrhage (sICH) transformation was defined according to European Cooperative Acute Stroke Study (ECASS)-III criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gang Li, Principal Investigator — Shanghai East Hospital
Locations (1):
- Gang Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarraj A, Hassan A, Savitz SI, Grotta JC, Cai C, Parsha KN, Farrell CM, Imam B, Sitton CW, Reddy ST, Kamal H, Goyal N, Elijovich L, Reishus K, Krishnan R, Sangha N, Wu A, Costa R, Malik R, Mir O, Hasan R, Snodgrass LM, Requena M, Graybeal D, Abraham M, Chen M, McCullough LD, Ribo M. Endovascular Thrombectomy for Mild Strokes: How Low Should We Go? Stroke. 2018 Oct;49(10):2398-2405. doi: 10.1161/STROKEAHA.118.022114. PMID 30355094
- [Result] Dargazanli C, Consoli A, Gory B, Blanc R, Labreuche J, Preda C, Bourdain F, Decroix JP, Redjem H, Ciccio G, Mazighi M, Smajda S, Desilles JP, Riva R, Labeyrie PE, Coskun O, Rodesch G, Turjman F, Piotin M, Lapergue B; ETIS investigators. Is Reperfusion Useful in Ischaemic Stroke Patients Presenting with a Low National Institutes of Health Stroke Scale and a Proximal Large Vessel Occlusion of the Anterior Circulation? Cerebrovasc Dis. 2017;43(5-6):305-312. doi: 10.1159/000468995. Epub 2017 Apr 7. PMID 28384632
- [Result] Shang X, Lin M, Zhang S, Li S, Guo Y, Wang W, Zhang M, Wan Y, Zhou Z, Zi W, Liu X. Clinical Outcomes of Endovascular Treatment within 24 Hours in Patients with Mild Ischemic Stroke and Perfusion Imaging Selection. AJNR Am J Neuroradiol. 2018 Jun;39(6):1083-1087. doi: 10.3174/ajnr.A5644. Epub 2018 May 3. PMID 29724764
- [Result] Dargazanli C, Arquizan C, Gory B, Consoli A, Labreuche J, Redjem H, Eker O, Decroix JP, Corlobe A, Mourand I, Gaillard N, Ayrignac X, Charif M, Duhamel A, Labeyrie PE, Riquelme C, Ciccio G, Smajda S, Desilles JP, Gascou G, Lefevre PH, Mantilla-Garcia D, Cagnazzo F, Coskun O, Mazighi M, Riva R, Bourdain F, Labauge P, Rodesch G, Obadia M, Bonafe A, Turjman F, Costalat V, Piotin M, Blanc R, Lapergue B; ETIS REGISTRY Investigators. Mechanical Thrombectomy for Minor and Mild Stroke Patients Harboring Large Vessel Occlusion in the Anterior Circulation: A Multicenter Cohort Study. Stroke. 2017 Dec;48(12):3274-3281. doi: 10.1161/STROKEAHA.117.018113. Epub 2017 Oct 31. PMID 29089458
- [Result] Haussen DC, Lima FO, Bouslama M, Grossberg JA, Silva GS, Lev MH, Furie K, Koroshetz W, Frankel MR, Nogueira RG. Thrombectomy versus medical management for large vessel occlusion strokes with minimal symptoms: an analysis from STOPStroke and GESTOR cohorts. J Neurointerv Surg. 2018 Apr;10(4):325-329. doi: 10.1136/neurintsurg-2017-013243. Epub 2017 Aug 2. PMID 28768820
- [Result] Kaesmacher J, Chaloulos-Iakovidis P, Panos L, Mordasini P, Heldner MR, Kurmann CC, Michel P, Hajdu SD, Ribo M, Requena M, Maegerlein C, Friedrich B, Costalat V, Benali A, Pierot L, Gawlitza M, Schaafsma J, Pereira VM, Gralla J, Fischer U. Clinical effect of successful reperfusion in patients presenting with NIHSS < 8: data from the BEYOND-SWIFT registry. J Neurol. 2019 Mar;266(3):598-608. doi: 10.1007/s00415-018-09172-1. Epub 2019 Jan 8. PMID 30617997
- [Derived] Liu F, Shen H, Chen C, Bao H, Zuo L, Xu X, Yang Y, Cochrane A, Xiao Y, Li G. Mechanical Thrombectomy for Acute Stroke Due to Large-Vessel Occlusion Presenting With Mild Symptoms. Front Neurol. 2021 Oct 28;12:739267. doi: 10.3389/fneur.2021.739267. eCollection 2021. PMID 34777207